CLINICAL TRIAL: NCT02185469
Title: Corneal Endothelial Cell Loss After Pneumatic Retinopexy for the Repair of Primary Rhegmatogenous Retinal Detachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Peter Kertes, Dr. Peter Kertes ,MD, CM, FRCSC Chief of Ophthalmology, Retina Specialist, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRECC001
Record Dates: First submitted 2014-06-09; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Corneal Endothelial Cell Loss; pneumatic retinopexy; vitrectomy
MeSH Terms: conditions — Corneal Endothelial Cell Loss | interventions — Vitrectomy; Sulfur Hexafluoride; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pneumatic retinopexy group (Active Comparator): First, a 5/8-in 25-gauge needle will be used to perform an anterior chamber paracentesis, aiming to withdraw a minimum of 0.3 ml of aqueous fluid form the anterior chamber. Then, sulfur hexafluoride (SF6) will be injected in the vitreous cavity. The total volume of gas injected will exceed by 0.3 ml the amount of fluid withdrawn by the anterior chamber paracentesis (ex: 0.6 ml of SF6 would be injected after having withdrawn 0.3 ml). The laser retinopexy will be performed 48 hours later with laser.
  Interventions: Procedure: Pneumatic retinopexy; Drug: sulfur hexafluoride (SF6); Device: 5/8-in 25-gauge needle; Device: laser
- vitrectomy group (Active Comparator): Under certain circumstances, pneumatic retinopexy can't be considered as a primary treatment for rhegmatogenous retinal detachment. In these cases, the patient will be booked for urgent 25 G vitrectomy with intraoperative laser retinopexy and gas injection to treat retinal detachment
  Interventions: Procedure: vitrectomy; Device: laser

INTERVENTIONS:
Procedure: Pneumatic retinopexy — First, a 5/8-in 25-gauge needle will be used to perform an anterior chamber paracentesis, aiming to withdraw a minimum of 0.3 ml of aqueous fluid form the anterior chamber. Then, sulfur hexafluoride (SF6) will be injected in the vitreous cavity. The total volume of gas injected will exceed by 0.3 ml the amount of fluid withdrawn by the anterior chamber paracentesis (ex: 0.6 ml of SF6 would be injected after having withdrawn 0.3 ml). The laser retinopexy will be performed 48 hours later with laser.
  Arms: pneumatic retinopexy group
Procedure: vitrectomy — Under certain circumstances, pneumatic retinopexy can't be considered as a primary treatment for rhegmatogenous retinal detachment. In these cases, the patient will be booked for urgent 25 G vitrectomy with intraoperative laser retinopexy and gas injection to treat retinal detachment
  Arms: vitrectomy group
Drug: sulfur hexafluoride (SF6)
  Arms: pneumatic retinopexy group
Device: 5/8-in 25-gauge needle
  Arms: pneumatic retinopexy group
Device: laser — intraoperative laser retinopexy

SUMMARY:
There are multiple ways to treat retinal detachment, the aim of this study is to compare the amount of corneal endothelial cell loss after pneumatic retinopexy in comparison to vitrectomy.

DETAILED DESCRIPTION:
Retinal detachment is a separation of the neurosensory retina from the retinal pigment epithelium. The most common form is rhegmatogenous retinal detachment, which occurs as the result of a full-thickness retinal break. There are three major techniques available to repair the detachment: scleral buckling, primary vitrectomy, and pneumatic retinopexy. At our institution, pneumatic retinopexy is the technique most commonly employed for primary repair. Pneumatic retinopexy is a minimally invasive surgery that involves injection of an intravitreal gas bubble to tamponade the causative retinal tear(s) and cryotherapy or laser photocoagulation to create a permanent chorioretinal adhesion.

Endothelial cells pumping function is essential to keep the cornea in a relatively dehydrated state that allows optical clarity. Corneal endothelial damage has been associated with almost all types of intraocular surgery. Cell loss due to vitrectomy in phakic eyes varies between 0.4 and 2.8%. , , , , During pars plana vitrectomy, all manipulation take place in the vitreous cavity; a certain distance from the corneal endothelium. Cataract extraction by phacoemulsification results in greater endothelial cell loss (4-18%), because of the greater proximity to the corneal endothelium during manipulation and direct damage from the use of ultrasound. To our knowledge, corneal endothelial cell loss after pneumatic retinopexy has never been studied. Corneal endothelium can be damaged during pneumatic retinopexy because an anterior paracentesis is performed before the gas injection. A 5/8-in 25-gauge needle is used to withdraw 0.3 to 0.35 ml of aqueous fluid form the anterior chamber. The procedure is invariably accompanied by a certain degree of shallowing of the anterior chamber. We postulate that endothelial cell damage can result from the direct contact of the needle tip with the corneal endothelium during wound creation and by inadvertent contact during shallowing of the anterior chamber.

A standard method of endothelial cell analysis used worldwide is specular microscopy. Specular microscopy is a non-invasive technique to access the structure and function of the corneal endothelium by permitting visualization of the corneal endothelial mosaic. From the areas of the cornea measured with specular microscopy, an estimate of endothelial cell density can be made.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* Patients with rhegmatogenous retinal detachment undergoing pneumatic retinopexy and pars plana vitrectomy.
* Patients on which specular microscopy and IOLMaster® can be performed without delaying their treatment (availability of a qualified operator).
* Decision makers able to give informed consent.

Exclusion Criteria:

* Unable to attend follow-up visits.
* History of previous intraocular surgery in surgical eye, except cataract extraction by phacoemulsification.
* Aphakia in surgical eye.
* Presence of an anterior chamber intraocular lens in surgical eye.
* Need for cryotherapy to treat the retinal break.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Endothelial cells count as measured by specular microscopy | at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kertes, MD, CM, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada